CLINICAL TRIAL: NCT00616265
Title: Effect of CPAP Treatment in the Control of Refractory Hypertension
Brief Title: Effect of Continuous Positive Airway Pressure (CPAP) Treatment in the Control of Refractory Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Principal Investigator, Miguel angel Martinez Garcia, MD, Sociedad Española de Neumología y Cirugía Torácica
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Prot-740; Prot-740 SEPAR; SEPAR-90 (Other: SEPAR)
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2012-02-29 (Estimated); Status verified 2012-02

CONDITIONS: Sleep Apnea; Hypertension
Keywords: Sleep apnea; Refractory Hypertension; Difficult-to-treat hypertension; CPAP
MeSH Terms: conditions — Sleep Apnea Syndromes; Hypertension | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- B (No Intervention): Group B. Only Usual Control
- A (Experimental): Group A: Cpap treatment plus Usual control
  Interventions: Device: CPAP

INTERVENTIONS:
Device: CPAP — Pressure device on airway to maintain it open
  Other Names: Continuous positive airway pressure
  Arms: A

SUMMARY:
The working hypothesis for the present study is that treatment with CPAP in patients with an sleep apnea (IAH>15) and AHT-r is capable of producing significant reductions in blood-pressure levels.

This hypothesis is supported by four proven findings:

1. -sleep apnea is an independent risk factor for arterial hypertension (1).
2. -The greater the number of RSD, the greater the loss of control over blood-pressure levels (1).
3. -The prevalence of sleep apnea in patients with AHT refractory to treatment is very high (11,12).
4. -Treatment of patients with sleep apnea and AHT-r with CPAP succeeds in significantly reducing blood-pressure levels in the only (small-scale) studies undertaken to date (14,15).

4. OBJECTIVES

Main objective:

To evaluate the effect of treatment with CPAP on blood-pressure levels in patients with AHT refractory to medical treatment.

Secondary objectives:

* To evaluate the effect of treatment with CPAP on the various elements assessed in BP (systolic/diastolic; daytime/nighttime, etc) and the circadian profile (dipper/non-dipper/raiser patterns; variability and homogeneity of blood-pressure levels, etc) obtained during a 24-hour out-patient study (AMPA).
* To analyze the related variables or subgroups of patients most affected by treatment with CPAP.
* To evaluate the effect of CPAP on the levels of some of the biological variables involved in the pathogenesis of AHT-r (renin, angiotensin, aldosterone, atrial natriuretic factor, etc).

DETAILED DESCRIPTION:
OBJECTIVE. To evaluate the effect of continuous positive airway pressure (CPAP) treatment on the blood-pressure (BP) levels of patients with refractory arterial hypertension (AHT-r).

METHODS: Multicenter randomized study with parallel groups and blind final evaluation.

Patients will be recruited from AHT, nephrology or internal medicine outpatient clinics and will satisfy the criteria for AHT-r (patients requiring 3 anti-AHT drugs at recommended doses to maintain their blood-pressure levels within AMPA [24-hours ambulatory monitoring of blood pressure values) excluding those forms of secondary AHT and those patients with incapacitating hypersomnia that need immediate treatment. In all, 210 patients will be included (105 per arm for intention to treat analysis) in accordance with the calculation of the sample size needed including drop-outs to evaluate a clinically significant minimum drop of 4-5 mmHg in the mean BP and the number of centers (21 centers; 10 patients per center). They will all be subjected to a complete clinical history, an AMPA study, a blood test (with serum retained for a later determination of biological mediators) and a sleep study. Those patients with an AHI>15 will be randomized to receive CPAP vs habitual control. The treatment will last 3 months. The same variables that were measured before the randomization will be analyzed again for the purposes of comparison. The comparison of results will be undertaken on the basis of an intention-to-treat and per-protocol analyses based on adherence to CPAP treatment at different cutoff of hours /day by means of an ANOVA two-way analysis (one of them being time).

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18-75 with a diagnosis of primary AHT-r and an AHI ≥15.
2. Signature indicating informed consent.

Exclusion Criteria:

1. Those patients with, in the opinion of the researcher, incapacitating hypersomnia will be excluded (to avoid the ethical problems associated with not treating a symptomatic sleep apnea patient).
2. Patients with risky professions or work involving dangerous goods.
3. Pregnancy.
4. The regular use of psychotropic drugs that could significantly modify the results of the sleep studies, or previous alcoholism (more than 100 gr of alcohol/day).
5. Patients previously treated with CPAP.
6. Record of poor compliance with anti-hypertensive treatment.
7. AHT secondary to cardiac insufficiency, valvulopathy, renal or endocrinological causes, cor pulmonale or the consumption of oral corticoids, or any other known cause.
8. Patients who have suffered from a cardiovascular event in the month prior to inclusion in the study, or patients who were unstable at the time of their inclusion in the study.
9. Known renal insufficiency with a concentration of creatinine greater than 1.5 mg/dl

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2008-06; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Effect on blood pressure levels | Before and six months after CPAP treatment

SECONDARY OUTCOMES:
Effect on night blood pressure pattern | Befor and six month after CPAP treatment

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Angel Martínez-Garcia, MD, Principal Investigator — Sociedad Española de Neumología y Cirugía Torácica
Locations (1):
- General Hospital of Requena, Valencia, Valencia, Spain

REFERENCES:
- [Derived] Sanchez-de-la-Torre M, Khalyfa A, Sanchez-de-la-Torre A, Martinez-Alonso M, Martinez-Garcia MA, Barcelo A, Lloberes P, Campos-Rodriguez F, Capote F, Diaz-de-Atauri MJ, Somoza M, Gonzalez M, Masa JF, Gozal D, Barbe F; Spanish Sleep Network. Precision Medicine in Patients With Resistant Hypertension and Obstructive Sleep Apnea: Blood Pressure Response to Continuous Positive Airway Pressure Treatment. J Am Coll Cardiol. 2015 Sep 1;66(9):1023-32. doi: 10.1016/j.jacc.2015.06.1315. PMID 26314530
- [Derived] Martinez-Garcia MA, Capote F, Campos-Rodriguez F, Lloberes P, Diaz de Atauri MJ, Somoza M, Masa JF, Gonzalez M, Sacristan L, Barbe F, Duran-Cantolla J, Aizpuru F, Manas E, Barreiro B, Mosteiro M, Cebrian JJ, de la Pena M, Garcia-Rio F, Maimo A, Zapater J, Hernandez C, Grau SanMarti N, Montserrat JM; Spanish Sleep Network. Effect of CPAP on blood pressure in patients with obstructive sleep apnea and resistant hypertension: the HIPARCO randomized clinical trial. JAMA. 2013 Dec 11;310(22):2407-15. doi: 10.1001/jama.2013.281250. PMID 24327037